CLINICAL TRIAL: NCT02604368
Title: A Phase 3, Prospective, Randomized, Double-Blind, Placebo Controlled, Multi-center Study of SC411 for Sickle Cell Disease
Brief Title: A Sickle CEll Disease ComplicatioN Trial
Acronym: ASCENT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Micelle BioPharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OMEG-411-01
Record Dates: First submitted 2015-11-11; First posted 2015-11-13 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Sickle Cell Disease
Keywords: hemoglobin SS; hemoglobin SC; hemoglobin S/β°-thalassemia
MeSH Terms: conditions — Anemia, Sickle Cell; Hemoglobin SC Disease | interventions — Docosahexaenoic Acids; Soybean Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SC411 (Experimental): Omega-3 docosahexaenoic acid, soft gelatin capsule, administered once a day on a per weight basis.
  Interventions: Drug: SC411
- Placebo (Placebo Comparator): Soybean oil, soft gelatin capsule, administered once a day on a per weight basis.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SC411 — Soft gelatin capsule
  Other Names: Docosahexaenoic acid (DHA)
  Arms: SC411
Drug: Placebo — Soft gelatin capsule
  Other Names: Soybean Oil
  Arms: Placebo

SUMMARY:
The objective of this study is to assess the efficacy of SC411 in reducing the number of sickle cell crisis (SCC) events in sickle cell disease (SCD) subjects receiving SC411 compared to those subjects receiving placebo.

DETAILED DESCRIPTION:
This Phase 3, prospective, randomized, double-blinded, placebo-controlled, multi-center study will enroll approximately 210 subjects at up to 70 sites in the United States. Participation will consist of a Screening Period, followed by a minimum 12-month Treatment Period. SC411 is administered orally as a soft gel mini capsule.

This study will enroll subjects aged ≥5 to ≤17 years who have a diagnosis of SCD that includes the phenotypes hemoglobin SS homozygous (HbSS), hemoglobin SC (HbSC), and hemoglobin S/β°-thalassemia (HbS/ β°-thalassemia); and have had at least 2 but no more than 10 documented SCC events (as defined above) within 12 months prior to the Screening Visit.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all of the following criteria will be eligible to participate in the study:

1. 1. Aged ≥ 5 years and ≤ 17 years at screening;
2. Has been diagnosed with SCD (that includes the genotypes HbSS, HbSC, and HbS/β°-thalassemia, documented by hemoglobin HPLC or electrophoresis);
3. Has had between ≥ 2 to ≤10 episodes of acute SCC (as defined above) within 12 months of the Screening Visit. At least one crisis must have been managed in a hospital, clinic, or emergency room. For at least 2 of the episodes, the site must obtain the documentation created in a medical record at the time of the event.
4. Must not be receiving HU or L-Glutamine, or if receiving HU and/or L-Glutamine must be at a stable weight-based treatment regimen (mg/kg), for at least 3 months prior to the Screening Visit with the intent to continue at a weight-based dose level at the discretion of the treating physician for the duration of the study, other than for safety reasons. If taking HU and/or L-glutamine, subjects must have had at least one SCC event (as previously defined) while on HU and/or L-Glutamine.
5. Has a parent or guardian who is able to give written informed consent, and the potential pediatric subject must be able to provide assent in a manner approved by the Institutional Review Board (IRB) and comply with the requirements of the study; and
6. If post pubertal in the opinion of the Investigator, must agree to use a reliable method of birth control (e.g., barrier, birth control pills, abstinence) during the study and for 1 month following the last dose of study drug.

Exclusion Criteria

Patients who meet any of the following criteria will be excluded from participation in the study:

1. A known allergy or hypersensitivity to fish or shellfish;
2. A known allergy or hypersensitivity to soy;
3. Inability to swallow capsules;
4. History of treatment with SC411;
5. Confirmed diagnosis of chronic pain or chronic opioid use: Defined as pain experienced ≥3 days per week over a 6-month period or daily opioid use for pain management;
6. Active infection with Human Immunodeficiency Virus (HIV), Hepatitis B, or Hepatitis C;
7. Prothrombin time > 1.5 x ULN at screening;
8. Required regular anticoagulation or chronic aspirin therapy;
9. Moderate thrombocytopenia, defined as platelets < 80,000/µL at screening;
10. History of stroke or Moyamoya syndrome;
11. Abnormal results on most recent transcranial Doppler (TCD) evaluation;
12. Received blood transfusion or blood products in the 2 months prior to the Screening Visit or on chronic blood transfusion;
13. Chronic renal insufficiency, defined as a eGFR < 30ml/min at screening as estimated by the Schwartz equation (Appendix H), or requiring peritoneal or hemodialysis;
14. Abnormal liver function tests (ALT > 3.0 x ULN) at screening;
15. Received any organ transplant;
16. Has a recent acute illness or other concomitant chronic medical or psychiatric condition that in the opinion of the Investigator would compromise participation in the study, prevent adherence to the protocol or confound the evaluation of the study outcome;
17. Is pregnant or lactating, or has the intention of becoming pregnant during the study (if a female of child-bearing potential or partner of a female of child-bearing potential and sexually active and not willing to use an effective means of birth control);
18. Is currently taking or has been treated with any form of omega-3 fatty acid or fish oil supplement within 30 days of the Screening Visit, or intends to do so during the course of the study;
19. Has been treated with any investigational product within 30 days of the Screening Visit or intends to receive an investigational product during the course of this study; and
20. There are factors that, in the judgment of the Investigator, would make it difficult for the patient to comply with the requirements of the study

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 210 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of the efficacy of SC411 in reducing the number of sickle cell crisis (SCC) events in subjects compared to placebo will be measured by counting the number of sickle cell crises that occur after randomization. | 52 weeks
  Assessment of the efficacy of SC411 in reducing the number of sickle cell crisis (SCC) events in subjects compared to placebo will be measured by counting the number of sickle cell crises that occur after randomization.
  The primary objective of this study is to assess the efficacy of orally administered SC411 in reducing the number of sickle cell crisis (SCC) events in sickle cell disease (SCD) subjects compared to placebo. A SCC event will be defined as either an acute painful crisis or an acute chest syndrome.

SECONDARY OUTCOMES:
Evaluation of the effect of SC411 compared to placebo by measuring the time until the patient's first sickle cell event. | 52 weeks
  Evaluation of days to the first event from randomization for each patient.
Evaluation of the effect of SC411 compared to placebo by measuring the the number of visits to a medical facility (hospital, clinic, or emergency room) for SCC event or complications of SCD. | 52 weeks
  Evaluation of the effect of SC411 compared to placebo by measuring the the number of visits to a medical facility (hospital, clinic, or emergency room) for SCC event or complications of SCD.
Evaluation of the effect of SC411 compared to placebo by measuring the number of days with electronic diary (eDiary)-recorded opioid or non opioid analgesic use at home to manage sickle cell pain. | 52 weeks
  To evaluate the effect of SC411 compared to placebo by measuring the number of days with electronic diary (eDiary)-recorded opioid or non opioid analgesic use at home to manage sickle cell pain.
Evaluation of the effect of SC411 compared to placebo by measuring the number of crisis-free days. | 52 weeks
  To evaluate the effect of SC411 compared to placebo by measuring the number of crisis-free days. A crisis-free day is defined as any day with a zero entry on the eDiary pain intensity scale.

OTHER OUTCOMES:
Evaluation of the effect of SC411 compared to placebo by measuring the time to second SCC event among subjects who had experienced at least one crisis while enrolled in the study. | 52 weeks
  To evaluate the effect of SC411 compared to placebo by measuring the time to second SCC event among subjects who had experienced at least one crisis while enrolled in the study.
Evaluation of the effect of SC411 compared to placebo by measuring the number of complications of SCD. | 52 weeks
  To evaluate the effect of SC411 compared to placebo by measuring the number of complications of SCD.
Evaluation of the effect of SC411 compared to placebo by measuring the Parent/guardian eDiary-recorded school attendance. | 52 weeks
  To evaluate the effect of SC411 compared to placebo by measuring the Parent/guardian eDiary-recorded school attendance.
Evaluation of the effect of SC411 compared to placebo by measuring the percent of days free of eDiary-recorded sickle cell pain out of total number of Treatment Period days. | 52 weeks
  To evaluate the effect of SC411 compared to placebo by measuring the percent of days free of eDiary-recorded sickle cell pain out of total number of Treatment Period days.
Evaluation of the effect of SC411 compared to placebo by measuring the subjects eDiary-recorded sickle cell pain score on the days that pain is recorded analyzed over time for intensity and diminution. | 52 weeks
  To evaluate the effect of SC411 compared to placebo by measuring the subjects eDiary-recorded sickle cell pain score (scale from 0-10) on the days that pain is recorded analyzed over time for intensity and diminution.
Evaluation of the effect of SC411 compared to placebo by measuring the subjects eDiary-recorded sickle cell pain score on the days during a SCC event analyzed over time for intensity and diminution. | 52 weeks
  To evaluate the effect of SC411 compared to placebo by measuring the subjects eDiary-recorded sickle cell pain score (from 0-10) on the days during a SCC event analyzed over time for intensity and diminution.
Evaluation of the effect of SC411 compared to placebo by measuring the number of hospitalization days due to SCC events. | 52 weeks
  To evaluate the effect of SC411 compared to placebo by measuring the number of hospitalization days due to SCC events.
  -
Evaluation of the effect of SC411 compared to placebo by measuring the number of hospitalizations due to SCC events. | 52 weeks
  To evaluate the effect of SC411 compared to placebo by measuring the number of hospitalizations due to SCC events.
Evaluation of the effect of SC411 compared to placebo by measuring the number of acute painful crisis events. | 52 weeks
  To evaluate the effect of SC411 compared to placebo by measuring the number of acute painful crisis events.
Evaluation of the effect of SC411 compared to placebo by measuring the number of acute chest syndrome events. | 52 weeks
  To evaluate the effect of SC411 compared to placebo by measuring the number of acute chest syndrome events.
Evaluation of the effect of SC411 compared to placebo by measuring the number of simple and exchange blood transfusions. | 52 weeks
  To evaluate the effect of SC411 compared to placebo by measuring the number of simple and exchange blood transfusions.
Evaluation of the effect of SC411 compared to placebo by measuring the changes in hemoglobin. | 52 weeks
  To evaluate the effect of SC411 compared to placebo by measuring the changes in hemoglobin.
Evaluation of the effect of SC411 compared to placebo by measuring the changes in hematocrit. | 52 weeks
  To evaluate the effect of SC411 compared to placebo by measuring the changes in hematocrit.
Evaluation of the effect of SC411 compared to placebo by measuring the changes in hemoglobin phenotype. | 52 weeks
  To evaluate the effect of SC411 compared to placebo by measuring the changes in hemoglobin phenotype.
Evaluation of the effect of SC411 compared to placebo by measuring the changes in white blood cells. | 52 weeks
  To evaluate the effect of SC411 compared to placebo by measuring the changes in white blood cells.
Evaluation of the effect of SC411 compared to placebo by measuring the changes in blood platelets. | 52 weeks
  To evaluate the effect of SC411 compared to placebo by measuring the changes in blood platelets.
Evaluation of the effect of SC411 compared to placebo by measuring the changes in the RBC membrane omega-3 fatty acids index. | 52 weeks
  To evaluate the effect of SC411 compared to placebo by measuring the changes in the RBC membrane omega-3 fatty acids index (arachidonic acid, docosahexaenoic acid, and eicosapentaenoic acid).
Evaluation of the effect of SC411 compared to placebo by measuring the changes in the reticulocyte count. | 52 weeks
  To evaluate the effect of SC411 compared to placebo by measuring the changes in the reticulocyte count.
Evaluation of the effect of SC411 compared to placebo by measuring the changes in lactate dehydrogenase. | 52 weeks
  To evaluate the effect of SC411 compared to placebo by measuring the changes in lactate dehydrogenase.
Evaluation of the effect of SC411 compared to placebo by measuring the changes in haptoglobin. | 52 weeks
  To evaluate the effect of SC411 compared to placebo by measuring the changes in haptoglobin.
Evaluation of the effect of SC411 compared to placebo by measuring the changes in indirect bilirubin. | 52 weeks
  To evaluate the effect of SC411 compared to placebo by measuring the changes in indirect bilirubin.
Evaluation of the effect of SC411 compared to placebo by measuring the changes in high sensitivity C-reactive protein. | 52 weeks
  To evaluate the effect of SC411 compared to placebo by measuring the changes in high sensitivity C-reactive protein.
Evaluation of the effect of SC411 compared to placebo by measuring the changes in D-dimer. | 52 weeks
  To evaluate the effect of SC411 compared to placebo by measuring the changes in D-dimer.
Evaluation of the effect of SC411 compared to placebo by measuring the changes in whole blood adhesion to vascular cell adhesion molecule-1. | 52 weeks
  To evaluate the effect of SC411 compared to placebo by measuring the changes in whole blood adhesion to vascular cell adhesion molecule-1.
Evaluation of the effect of SC411 compared to placebo by measuring the changes in E-selectin. | 52 weeks
  To evaluate the effect of SC411 compared to placebo by measuring the changes in E-selectin.

CONTACTS AND LOCATIONS:
Overall Officials: Carton Dampier, MD, Study Chair — Emory University; Matt Heeney, MD, Study Chair — Harvard University; Beng Fuh, MD, Study Chair — East Carolina University